CLINICAL TRIAL: NCT06728280
Title: Efficacy and Safety of Deep Transcranial Magnetic Stimulation in Adolescent Major Depressive Disorder: a Prospective Double-Blind Randomized Controlled Trial
Brief Title: Efficacy and Safety of DTMS in Adolescent Major Depressive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhifen Liu (Other)
Responsible Party: Sponsor-Investigator, Zhifen Liu, professor, The First Affiliated Hospital of Shanxi Medical University
Organization: The First Affiliated Hospital of Shanxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NO.KYLL-2024-001
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Diorder
Keywords: deep transcranial magnetic stimulation; Major Depressive Diorder; adolescents

STUDY DESIGN:
Intervention Model Description: randomized, double-blind,single-center, two-arm, parallel-group superiority trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Given the study's design, blinding TMS operators will not be possible. Still, participants、staff responsible for participant assessments and data analysis will be blinded to treatment conditions and external to the clinic staff. Patients will be instructed not to reveal their group assignment to the raters. Patients will not be given the specifics of the treatment parameters and will be instructed not to talk to each other during the study period. Both treatments will be presented as effective to them. Lastly, the data management center will strictly control access to the randomization code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- H1 coil (Active Comparator): First, the 'hot spot' for activation of the abductor pollicis brevis muscle was established and motor threshold (MT) determined. Then, the H1 coil was advanced 6 cm anterior to the scalp surface.The rMT was rechecked at least once a week. Treatment intensity was 80% of rMT.During 4 consecutive weeks (5 sessions/wk) patients were treated daily . Patients in the treatment group will receive the Deep TMS protocol (80% of rMT, 18 Hz, 2 seconds on and 20 seconds off over a 20-minute period; total of 1,980 stimuli per session), applied over the left dorsolateral prefrontal cortex.
  Interventions: Device: deep transcranial magnetic stimulation with H1coil
- H7 coil (Experimental): First, the 'hot spot' for activation of the abductor pollicis brevis muscle was established and motor threshold (MT) determined. Then, the H7 coil was advanced 4 cm anterior to 'hot spot' and aligned symmetrically over the dmPFC. The rMT was rechecked at least once a week.The rMT was rechecked at least once a week. Treatment intensity was 80% of rMT.During 4 consecutive weeks (5 sessions/wk) patients were treated daily . Patients in the treatment group will receive the Deep TMS protocol (80% of rMT, 18 Hz, 2 seconds on and 20 seconds off over a 20-minute period; total of 1,980 stimuli per session), applied over themedial prefrontal cortex.
  Interventions: Device: deep transcranial magnetic stimulation with H7 coil

INTERVENTIONS:
Device: deep transcranial magnetic stimulation with H1coil — Participants will receive dTMS treatment with H1 coil
  Arms: H1 coil
Device: deep transcranial magnetic stimulation with H7 coil — Participants will receive dTMS treatment with H7 coil
  Arms: H7 coil

SUMMARY:
The goal of this randomized controlled trial is to explore the efficacy and safety of two different dTMS devices in adolescent depression: deep TMS H1 coil and deep TMS H7 coil.

The main questions it aims to answer are:

Type of study: Clinical trial. Participant population: Adolescents with major depressive disorder (MDD). Objective: To explore whether the H7 coil is no less effective than the H1 coil for adolescents with MDD, further providing clinicians with additional treatment options for patients.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a safe and well-tolerated intervention that has been extensively studied as a treatment for MDD. However, little is known about the effectiveness of deep transcranial magnetic stimulation (dTMS) in adolescents with major depressive disorder (MDD). Only one open-label trial tested dTMS using H1 coils in adolescents with treatment-resistant depression, the results showed that the severity of depressive symptoms was significantly reduced after treatment, with a response rate of 42%. Hence, the continued efforts are needed to improve and optimize these treatments.

One important factor that influence the efficacy of TMS was the seletion of stimulation target. In recent years, medial prefrontal cortex (MPFC) and anterior cingulate cortex (ACC) have recently been considered promising alternative targets for treatment of adolescents with MDD, due to their association with reward, emotion, mood, and habits. Additionally, the stimulation target for dTMS with the H7 coil is the MPFC. Current relevant clinical studies show that after dTMS intervention using the H7 coil, depressive symptoms and overall clinical impressions in adults with MDD are significantly improved. However, whether alternative strategies for TMS treatment (e.g., H1 coil versus H7 coil) are more effective in adolescents with MDD remains unknown.

The purpose of this randomized controlled trial is to evaluate the efficacy and safety of two different dTMS devices (H1 coil and H7 coil) in the treatment of adolescent with MDD, further providing clinicians with additional treatment options for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders, aged between 11 and 23 years old, and right-handedness.
* In accordance with the diagnostic criteria for the major depressive disorder of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
* The current major depressive episode (MDE) must be confirmed using the Mini International Neuropsychiatric Interview (M.I.N.I).
* Beck Depression Inventory, Second Edition (BDI-II): total BDI-II score> 13 at screening.
* Subjects who can understand and are willing to strictly follow the clinical trial protocol to complete this study and sign informed consent.

Exclusion Criteria:

* A diagnosis of other psychiatric disorders in the DSM-5.
* Clinically significant laboratory abnormality or medical condition, that in the opinion of the investigator would hinder the subject in completing the procedures required by the study.
* History of significant neurologic disease, including subdural hematoma, brain tumor, unexpected seizure/epilepsy disorder, or history of significant head trauma.
* Have obvious suicide risk, or have actual suicide behavior within 6 months before the screening.
* History of treatment with electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), transcranial Direct Current Stimulation (tDCS), or transcranial Alternating Current Stimulation (tACS) treatments for any disorders.
* There are contraindications to magnetic resonance imaging (MRI) scanning or TMS treatment, such as metal or electronic instruments.
* Participation in any investigational drug trial within 6 months before the baseline visit.
* Other conditions that are not suitable for the study object in the researcher's judgment.

Ages: 11 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale -24 (HAMD-24) | From enrollment to the end of treatment at 12 weeks
  score change. Higher score means worse outcome.(Min = 0, Max = 76)
Response on Hamilton Depression Scale-24 | From enrollment to the end of treatment at 12 weeks
  Defined as a score reduction of 50% or more
Remission onHamilton Depression Scale-24 | From enrollment to the end of treatment at 12 weeks
  Defined as a score of 7 or less

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | From enrollment to the end of treatment at 12 weeks
  score change. Higher score means worse outcome.(Min = 0, Max = 56)
Snaith-Hamilton Pleasure Scale (SHAPS) | From enrollment to the end of treatment at 12 weeks
  score change. Higher score means worse outcome.(Min= 0, Max = 56)
Beck Scale for Suicide Ideation-Chinese Version (BSI-CV) | From enrollment to the end of treatment at 12 weeks
  score change. Higher score means worse outcome.(Min= 0, Max = 38)
Self-Injury Diary Card | From enrollment to the end of treatment at 12 weeks
  Higher numeric value means worse outcome.
Pittsburgh sleep quality index(PSQI) | From enrollment to the end of treatment at 12 weeks
  Higher score means worse outcome.(Min= 0, Max = 21)
Clinical Global Impression (CGI) | From enrollment to the end of treatment at 12 weeks
  Higher score means worse outcome.(Min= 0, Max = 7)
Repeatable Battery for the Assessmental of Neuropsychological Status(RBANS) | From enrollment to the end of treatment at 12 weeks
  Lower score means worse outcome.(Min=40, Max = 160)
Brief Symptom Inventory-18(BSI-18) | From enrollment to the end of treatment at 12 weeks
  Higher score means worse outcome.(Min= 0, Max = 90)
Beck Depression Inventory-II | From enrollment to the end of treatment at 12 weeks
  score change. Higher score means worse outcome.(Min= 0, Max = 63)

CONTACTS AND LOCATIONS:
Locations (1):
- Deep Transcranial Magnetic Stimulation, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No